CLINICAL TRIAL: NCT02707679
Title: Comparison of Short-Term Effects of Mobilization With Movement and Kinesiotaping on Pain, Function and Balance in Patellofemoral Pain Syndrome: A Randomized Control
Brief Title: Comparison of Effects of Mobilization With Movement and Kinesiotaping in Patellofemoral Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, SERDAR DEMIRCI, Research Asistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LUT 12/175
Record Dates: First submitted 2016-03-02; First posted 2016-03-14 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: Knee; Mobilization; Taping; Function; Balance
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Traction; Movement; Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Effects of Mulligan's Mobilization (Other): The patients in this arm (n=18) received two techniques pertaining to Mulligan's Mobilization with movement approach (Mulligan's Straight Leg-Raise with Traction and Tibial Gliding) along with an exercise therapy. Patients received 4 sessions of treatment twice a week for a period of 2 weeks and followed up in accordance with a 6-week-home exercise program. Primary outcomes: pain severity, knee range of motion, hamstring flexibility, and physical performance (10-step stair climbing test, timed up and go test), Kujala Patellofemoral Pain Scoring and Y-Balance test were assessed before the treatment, 45 minutes after the initial treatment, at the end of the 4-session-treatment during 2-week period and 6 weeks later.
  Interventions: Other: Mulligan's Straight leg-raise with traction; Other: Mulligan's Mobilization with Movement; Other: Exercise
- Effects of Kinesiotaping (Other): Patients in this arm were applied kinesiotaping on quadriceps and hamstring muscle along with an exercise therapy. Patients received 4 sessions of treatment twice a week for a period of 2 weeks and followed up in accordance with a 6-week-home exercise program. The same assessment parameters was conducted on this arm too.
  Interventions: Other: Kinesiotaping; Other: Exercise

INTERVENTIONS:
Other: Mulligan's Straight leg-raise with traction — Mulligan's Straight leg raise technique was performed on patients with patellofemoral pain syndrome. The extremity on which the practice would be performed in supine position was grasped from the ankle level and was, then, subjected to traction longitudinally. Afterwards, the knee was lifted up passively while in extension and was kept for waiting for a few seconds at the point where tension was felt and was, then, returned to its initial position. The practice was repeated 10 times, and 3 sets of practice at 1-minute-intervals were performed.
  Arms: Effects of Mulligan's Mobilization
Other: Mulligan's Mobilization with Movement — Mulligan's Mobilization with Movement technique was performed on patients with patellofemoral pain syndrome. Each patient was tested in every direction in the course of the active knee flexion-extension movement so as to find out the best pain-free tibial gliding direction (medial-lateral part of the tibia, anterior-posterior, internal-external rotation). At the time of the active movement of the knee, the tibial gliding direction where pain was felt at the least was selected as the treatment direction of mobilization technique along with movement. The practice was performed by doing 10 repetitions for 3 sets and by providing 1-minute-resting time between the sets.
  Arms: Effects of Mulligan's Mobilization
Other: Kinesiotaping — Kinesiotaping was applied on patient with patellofemoral pain syndrome. To maintain proprioceptive stimulation in the quadriceps (from origo towards insertio) and to alleviate the tension of hamstring muscle, a 'Y''-shaped kinesiotape was applied by using the muscle technique.
  Arms: Effects of Kinesiotaping
Other: Exercise — All the patients were provided with several exercises within the scope of the home exercise program, such as hamstring muscle stretching, quadriceps isometric exercises, 4-way-strengthening with exercise elastic bands for the muscles of the hip, knee locking on foot and mini-squatting exercises. They were asked to do these exercises in 3 sets a day along with 10 repetitions for a period of 6 weeks.

SUMMARY:
Patellofemoral Pain Syndrome (PFPS), also known as the anterior knee pain, is one of the most common musculoskeletal disorders. Most of the patients suffer from knee pain for long time. The aim of this study was to investigate the short-term effects of Mobilization with movement and Kinesiotaping on pain, function and balance in patient with PFPS.

DETAILED DESCRIPTION:
Patellofemoral Pain Syndrome is one of the most common musculoskeletal problem in the world. It's incidence is also becoming higher and most people who have knee pain suffer from it for long time. In the treatment of PFPS, conservative treatment methods are preferred prior to surgical ones. When the literature was reviewed, no study in which Mobilization with movement (MWM) method was used and in which the effects of it was shown and compared with (Kinesiotaping) KT has been found so far with respect to the treatment of PFPS. Thirty-five female patients diagnosed with unilateral PFPS were randomly assigned into 2 groups. The patients in the first group (n=18) received two techniques of Mobilization with movement intervention while Kinesiotaping was applied to the other group (n=17). Both groups were treated with exercise. All patients received 4 sessions of treatment twice a week for a period of 2 weeks and followed up in accordance with a 6-week-home exercise program. Primary outcomes: pain severity, knee range of motion, hamstring flexibility, and physical performance (10-step stair climbing test, timed up and go test), Kujala Patellofemoral Pain Scoring and Y-Balance test were assessed.

ELIGIBILITY:
Inclusion Criteria:

* having knee pain at least 3 months and more than 3 points according to visual analog scale

Exclusion Criteria:

* no complying to the rehabilitation
* if patient wants to finished and want to complete study, they were excluded
* having meniscus, bursa, ligament, patellar tendon lesions, patellofemoral dislocation and/or recurrent subluxation, undergone lower extremity surgery

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2013-05; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Knee pain measured with Visual Analog Scale | 6 weeks
  Patient's knee pain was measured with Visual Analog Scale

SECONDARY OUTCOMES:
Knee joint range of motion was measured Universal goniometer. | 6 weeks
  Universal goniometer was used for evaluating the knee joint range of motion.
Balance measured with Y- Balance Test | 6 weeks
  The dynamic balance measurements of the patients were evaluated through Y- Balance Test
Function was measured with 10-step-ascent & descent stair-climbing test. | 6 weeks
  To evaluate the functional performances of the patients, 10-step-ascent & descent stair-climbing test was used.
Function was measured Kujala patellofemoral scoring system | 6 weeks
  Patient's function was measured with Kujala patellofemoral scoring system
Function was measured with timed up&go test | 6 weeks
  To evaluate the functional performances of the patients, timed up&go test was used.
Hamstring muscle flexibility was measured Universal goniometer. | 6 weeks
  Universal goniometer was used for evaluating the hamstring muscle flexibility.

CONTACTS AND LOCATIONS:
Overall Officials: Volga Bayrakcı Tunay, Prof., Study Director — supervisor of the study

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Djordjevic OC, Vukicevic D, Katunac L, Jovic S. Mobilization with movement and kinesiotaping compared with a supervised exercise program for painful shoulder: results of a clinical trial. J Manipulative Physiol Ther. 2012 Jul;35(6):454-63. doi: 10.1016/j.jmpt.2012.07.006. Epub 2012 Aug 24. PMID 22921332
- [Result] Kuru T, Yaliman A, Dereli EE. Comparison of efficiency of Kinesio(R) taping and electrical stimulation in patients with patellofemoral pain syndrome. Acta Orthop Traumatol Turc. 2012;46(5):385-92. doi: 10.3944/aott.2012.2682. PMID 23268824
- [Result] Collado H, Fredericson M. Patellofemoral pain syndrome. Clin Sports Med. 2010 Jul;29(3):379-98. doi: 10.1016/j.csm.2010.03.012. PMID 20610028